CLINICAL TRIAL: NCT04626349
Title: International Randomized Controlled Trial to Evaluate the Effectiveness of a Nurse-delivered (FOCUS+) and a Web-based (iFOCUS) Psychoeducational Intervention for People With Advanced Cancer and Their Family Caregivers
Brief Title: International Study to Evaluate Two Programs of Support for Patients With Advanced Cancer and Their Families
Acronym: DIAdIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Erasmus Medical Center (Other); King's College London (Other); Queen's University, Belfast (Other); University Ghent (Other); University of Copenhagen (Other); University of Dublin, Trinity College (Other); University College Dublin (Other); Azienda USL di Reggio Emilia (Unknown); European Commission (Other)
Responsible Party: Principal Investigator, Joachim Cohen, Professor of Public Health and Palliative Care, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EU grant agreement No 825722
Record Dates: First submitted 2020-10-27; First posted 2020-11-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Advanced Cancer
Keywords: psychoeducational intervention; quality of life; self-efficacy; randomized clinical trial; oncology; family caregiver
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Masking Description: Due to the nature of the intervention neither the patient-caregiver dyads nor the intervention nurses (for the face-to-face FOCUS+ intervention) can be blinded to allocation. Data will be collected via a computer-assisted self-interview with a data collector that is present for assistance and additional explanations. Those conducting the data analyses will be unaware as to what trial arm dyads were randomized to until the end of the last data collection point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FOCUS+ (Experimental): Dyads in the FOCUS+ arm will receive the face-to-face nurse-led FOCUS+ program.
  Interventions: Other: FOCUS+ (face-to-face nurse-led intervention)
- iFOCUS (Experimental): Dyads in the iFOCUS arm will receive the web-based iFOCUS program.
  Interventions: Other: iFOCUS (web-based intervention)
- Standard care (No Intervention): Dyads in the control group will receive standard care as usual, as determined by the healthcare system in the participating countries. The dose and frequency of usual care will be as deemed appropriate by the medical practitioner in charge of their treatment.

INTERVENTIONS:
Other: FOCUS+ (face-to-face nurse-led intervention) — Home-based psycho-educational intervention consisting of two 90-minute home visits and one 30-minute video-conferencing session, conducted by a trained intervention nurse over a period of 12 weeks (4 weeks between each session).
  The intervention is comprehensively manualized and there is a protocol to guide delivery of the intervention for each home visit and video call. The content of the sessions is always tailored to the needs of the dyads, so certain topics can be discussed more in-depth and specific information can be shared. The nurses who will deliver the FOCUS+ intervention will receive an extensive online training and additional continuous follow-up training to provide them with the knowledge and skills required to successfully implement the intervention. A FOCUS+ core booklet is provided as a supporting guide for the dyads that they can refer to at their own discretion and reinforces key intervention messages linked to the core components of the intervention.
  Arms: FOCUS+
Other: iFOCUS (web-based intervention) — Self-managed psycho-educational intervention that is completed autonomously by the patient-caregiver dyads together. It encompasses four sessions (with three weeks between each session) over a period of 12 weeks.
  The sessions are completed simultaneously by the patient and the family caregiver, sitting side by side at a computer. Patient-caregiver dyads have flexibility as to when they want to complete the intervention session. Based on the information patients and caregivers provided at enrollment and during the web-based sessions, they receive tailored individual and dyadic messages. An online personal workbook is provided containing the results of the interactive exercises that are provided to the dyads during the web-sessions. Any information brochures, leaflets and information sheets that the dyad indicated as 'of interest to them' during the web-sessions will be included as a hyperlink in their personal workbook.
  Arms: iFOCUS

SUMMARY:
The overall aim of this project is to evaluate the effectiveness, cost-effectiveness and mechanisms of action of two psychoeducational interventions (a face-to-face nurse-led intervention called FOCUS+ and an eHealth intervention called iFOCUS) aimed at improving the emotional function and self-efficacy of patients with advanced cancer and their family caregiver. Both interventions are compared to care as usual.

Both interventions focus on teaching dyads optimal ways to jointly manage the implications of advanced cancer and responding to their priority concerns and are designed to be tailored to the specific needs and wishes of the patient-caregiver dyads. Tailoring is based on information about the dyad obtained at enrollment (e.g. age, relationship, etc.) and the responses in the intervention sessions.

The overarching aim is addressed by five core intervention components:

1. supporting family involvement and improving the dyads mutual communication,
2. supporting outlook (i.e. increasing the dyad's capacity to identify positive or meaningful aspects related to their situation),
3. increasing dyads' coping skills, i.e. their capacity to identify their coping strategies and take action
4. help dyads reduce their uncertainty
5. teaching symptom management and giving them confidence to handle specific tasks and problems

Project objectives:

1. To compare 1) the face-to-face FOCUS+ intervention and 2) the iFOCUS web intervention to 3) care as usual in terms of their:

   * Effect on the emotional function and self-efficacy (primary outcomes), appraisal of illness, uncertainty, hopelessness, coping, dyad communication, quality of life and healthcare resource use of patients with advanced cancer and their family caregivers
   * Cost-effectiveness
   * Effects on vulnerable subgroups (particularly women and those of lower socioeconomic status)
   * Effectiveness in different healthcare systems
2. To evaluate the implementation process of the interventions in terms of the acceptability, feasibility, usefulness as perceived by patients, family caregivers and healthcare staff in each country, and their mechanisms of action.

Data will be collected three times from patient-caregiver dyads: 1) baseline measure (t0) after which the dyad will immediately be randomized to one of the study arms, 2) first follow-up at 12 weeks after baseline (t1) and 3) second follow-up at 24 weeks after baseline (t2).

DETAILED DESCRIPTION:
STUDY SETTING

Both interventions (FOCUS+ and iFOCUS) will be administered in the homes of the patient-caregiver dyads (or in the location of the dyad's preference).

The intervention will be conducted in six countries (Belgium, Denmark, Ireland, Italy, the Netherlands and the United Kingdom). In each country, patients with advanced cancer and their primary family caregiver will be recruited and enrolled via participating hospitals. Inclusion criteria for hospitals participating in this study are having 1) to treat patients with advanced cancer and 2) an oncology care regimen.

SAMPLE SIZE

For the emotional functioning the EF10 subscale from the EORTC is used. For self-efficacy the CASE instrument is used. The investigators consider demonstration of an intervention effect (for each of both interventions) on at least one of these primary outcomes for either the patient or the caregiver at t1 as a success. A pre-determined strict fixed sequence (FS) procedure defines prospectively hierarchical ordering of the endpoints, for this study the hierarchical order is emotional functioning (1) and self-efficacy (2). Testing of null hypotheses proceeds according to their hierarchical order, that is, H(1)0 is tested first at a significance level of 5%, and if H(1)0 is rejected then H(2)0 is tested at the same significance level, otherwise H(2)0 is not tested at all. The strict FS approach has the highest power for testing the first hypothesis (outcome: emotional function) compared to the other methods, as it does not save any portion of alpha for testing later hypothesis. The reference mean value from EORTC for all cancer patients, stage III-IV is 71.5 (SD: 23.8). Alpha is set at 0.0125 instead of 0.05 to account for multiplicity (2 comparisons with control group * 2 participant groups [patients and caregivers]). 1-beta (i.e. statistical power) is set at 0.9. The expected difference between the control group and the intervention arms in the primary outcomes is 0.375 SD at t1 (12 weeks).

With these parameters n= 203 is needed in each arm across all countries (i.e. 609 in total). Anticipating a 65% retention rate at t1, which is more conservative than found in previous studies in the USA on the FOCUS interventions due to the advanced cancer population included in this study, 938 dyads must be enrolled across the 6 countries (313 per group). This means n= 156 need to be enrolled in total in each country (n=52 in each of the 3 arms per country). Based on previous studies in the USA an enrolment rate of 55% is expected of those dyads referred to the study, meaning that about 282 dyads will need to be screened and identified in each country. The feasibility of recruitment has been evaluated based on previous research and discussions with clinicians in eligible hospitals.

DATA ANALYSIS

Four main quantitative analyses will take place:

1. Primary hypotheses testing:

   1. Testing the null hypothesis of the first primary endpoint: emotional functioning. The effectiveness of the FOCUS+ face-to-face intervention and the iFOCUS web-based intervention will be compared with the standard care (control group) for each participant population (patients/caregivers) separately. In total, 4 comparisons are performed for one outcome variable (alpha=0.0125). The hypotheses related to the first primary outcome (emotional functioning) will be tested using a mixed model (per participant population) with the T1 measurement value for emotional functioning as outcome variable, recruitment center as random effect and randomization group and baseline measure of emotional functioning (T0) as predictor variables. Analyses will be performed on both 'intention-to-treat' and per-protocol principles. The primary principle is intention-to-treat. After completion of the baseline measurement (T0), dyads will be randomized to one of the trial arms. All randomized dyads will be included in the mixed model. Multiple imputation will be applied. Predictors for the imputation model will include the baseline measurement, randomization group, age and other variables (e.g. severity of the illness). The secondary principle is the per-protocol analysis that functions as a sensitivity analysis. The per-protocol population will be defined as dyads who have completed all sessions of the FOCUS+ or iFOCUS intervention (except for dyads in the control group) and T1 measurement. By including the baseline measurement as a predictor variable (ANCOVA), preexisting differences will be controlled, enhancing the sensitivity of the analyses. To interpret the magnitude of the effects for the different outcomes, effect sizes (Cohen's d) will be estimated.
   2. Testing the null hypothesis of the second primary endpoint: self-efficacy (the Lewis´ Cancer self-efficacy scale from FOCUS) As per the fixed sequence (FS) procedure, the null hypotheses of the second primary endpoint (self-efficacy) will only be tested if a significant result is found for the first primary endpoint (emotional function). The same strategy is then followed for the analyses as for the first primary endpoint, with an alpha level of 0.0125.
2. Secondary hypotheses testing:

   All identified secondary endpoints (Quality of Life [including separate items of hopelessness, anxiety, depression], benefits of illness, coping, dyad communication, all at t1) will be evaluated by testing the FOCUS+ and iFOCUS will against care as usual (control group) for each participant population (patients/caregivers) separately. In total, 4 comparisons are performed for each outcome variable. For each secondary outcome variable a mixed model is applied (per participant population) with the T1 measurement value as outcome variable, recruitment center as random effect and randomization group and baseline measurement of the variable (T0) as predictor variables. Analyses will be performed on both 'intention-to-treat' and per-protocol principles, applying the same principles as described above.

   By including the baseline measurement as a predictor variable (ANCOVA), preexisting differences will be controlled, enhancing the sensitivity of the analyses. To interpret the magnitude of the effects for the different outcomes, effect sizes (Cohen's d) will be estimated. All statistical tests will be two-sided and considered significant if p< 0.0125.

   All primary outcomes and secondary outcomes as listed above will also be analysed at T2 (6 months) to evaluate longer term effects, using the same analysis procedures.

   The cost-effectiveness of the interventions will be determined by analyzing patterns and costs of healthcare utilization and effects on quality of life (measured by the EORTC, EQ5D5L, FACT G and CQOLC). Data will also be collected on the types and amounts of informal care provided to patients in each arm of the study, to investigate if amount or patterns of informal care change as a result of the intervention. The outputs will be mean costs of care for patients in each arm of the study, cost per year of life gained (if survival is affected significantly by the intervention and the costs in the intervention groups overall are higher) and (if appropriate) the additional costs of achieving better quality of life outcomes (including estimates of cost per quality adjusted life year gained).
3. Exploratory hypotheses testing:

   For all exploratory endpoints, two-sided statistical tests will be considered significant if p< 0.05
   1. For the outcomes that are measured identical for the patient and the caregiver, the effect on the dyad as a whole (i.e. both patient and family caregiver) will be assessed. For the outcome instruments that led to comparable estimated differences between FOCUS+ and standard care and iFOCUS and standard care, the effect will be assessed on the dyad as a whole by adding an extra level (dyad) to the linear regression model.
   2. For each of the primary and secondary endpoints, subgroup analyses will be performed using formal interaction tests to explore the extent to which the outcomes of the trial differ by country, gender and socioeconomic status. Interaction terms between respectively country, gender and socioeconomic status on the one hand and the trial arms on the other hand will be added to the analysis models. For the country variation a multilevel mixed model analyses will also be performed to additionally account for potential clustering by country (i.e. participants nested within a country). Outcomes will be analyzed with country as random factor.
4. Other analyses:

   1. Background reports describing care as usual for people with advanced cancer will facilitate the understanding of the results of the between-country comparisons.
   2. Process evaluation of the implementation of the interventions will be analyzed following the MRC framework for evaluating complex interventions, integrating normalization process theory (NPT) and the RE-AIM framework. Data analysis for the process evaluation will include a) standard statistical descriptions of the quantitative data from the intervention checklist and routine monitoring to describe adherence to the implementation. This analysis will determine cut-off points for good intervention adherence and, hence, inform the per-protocol analyses; b) analyses of the qualitative data (semi-structured interviews with patients and their family caregiver and post-intervention interviews with the nurses who delivered the face-to-face FOCUS+ intervention) will be performed (see below - Qualitative analysis).

Qualitative analysis:

With the transcription of interviews into the local language, the analysis process will involve a collaborative process involving researchers from each partner site collecting data. Thematic analysis allows for both inductive and deductive analysis and can be implemented with a range of computer-based software to support the management of the analysis process (e.g., NVIVO, MAXQDA).

Deductive analysis will be informed by semantic information sought from the interview (i.e., were participants satisfied, where particular elements of the programmes described as positive or negative) and themes evident in previous evaluations of the FOCUS intervention. This will involve developing themes in advance of the analysis process and assessing the presence or absence of these themes across the data. Inductive analysis will be structured using the objectives of the process evaluation to target key topics, with more latent or interpretative themes isolating more experiential findings from the data. Qualitative analysis will be conducted at two levels, an initial assessment of themes in each data source (stakeholders, staff, researchers, patients and carers, different language groups) followed by a higher-level analysis of superordinate themes of convergence and divergence evident across groups. Additional strategies for managing the potential impact of multilingual analysis are recommended, including peer debriefing during the process of coding and the development of candidate themes, triangulation across researchers and language sources. Analysis will be informed by open discussion of conceptual issues in the data to explore variations in interpretation and identify shared meaning relevant to the focus of the process evaluation.

ELIGIBILITY:
PATIENT

Inclusion Criteria:

* Diagnosis of cancer: solid organ (lung, colorectal, breast, prostate and other)
* No longer receives curative treatment (only life-prolonging or palliative treatments)
* Written informed consent
* Lives within feasible distance for intervention nurses to travel

Exclusion Criteria:

* Brain cancer, non-solid cancers
* Prognosis of less than 3 months
* Has no informal caregivers
* < 18 years old
* Unable to participate in available languages

FAMILY CAREGIVER

Inclusion Criteria:

* Written informed consent
* Primary informal caregiver as determined by the patient
* Lives within feasible distance for intervention nurses to travel

Exclusion Criteria:

* Unable to physically or mentally participate
* Cancer diagnosis in the last 12 months
* <18 years old
* Unable to participate in available languages

DYAD

Inclusion Criterium:

* Patient and/or family caregivers has access to and is familiar with use of internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in emotional functioning | T1 (baseline + 12 weeks)
  For patients and for caregivers: EORTC 10 emotional function items
Change in self-efficacy | T1 (baseline + 12 weeks)
  For patients and for caregivers: the Lewis´ Cancer self-efficacy scale

SECONDARY OUTCOMES:
Change in emotional functioning | T2 (baseline + 24 weeks)
  For patients and for caregivers: EORTC 10 emotional function items
Change in self-efficacy | T2 (baseline + 24 weeks)
  For patients and for caregivers: the Lewis´ Cancer self-efficacy scale
Change in patient quality of life | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients: EORTC QLQ-C15-PAL
Change in caregiver quality of life | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For caregivers: Caregiver Quality of Life Index-Cancer (CQOLC)
Change in patient social well-being | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients: social well-being scale from Functional Assessment of Cancer Therapy - General (FACT-G)
Change in patient social functioning | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients: 2 social functioning items from EORTC QLQ-C30
Change in patient overall health | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients: two items about overall health from EORTC QLQ-C30
Change in benefits of illness | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients and for caregivers: Benefits of illness scale
Change in coping | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients and for caregivers: A shortened version of Brief Cope
Change in ways of giving support | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients and for caregivers: The five items 'Active engagement scale' from the ´Ways of giving support questionnaire´.
Change in utilization of healthcare and associated services | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients and for caregivers: Client Service Receipt Inventory (CSRI)
Change in dyadic coping | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients and for caregivers: Three scales from the 'Dyadic Coping Inventory': 'Stress communication by oneself', 'Stress communication by partner' and 'Evaluation of dyadic coping'.
Change in quality-adjusted life years | T1 (baseline + 12 weeks), T2 (baseline + 24 weeks)
  For patients and for caregivers: EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Cohen, MSc, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (13):
- Belgium (4):
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Damiaan, Ostend
- Denmark (2):
  - Herlev University Hospital, Copenhagen
  - Rigshospitalet University Hospital, Copenhagen
- St. Vincent's University Hospital, Dublin, Ireland
- Azienda USL-IRCCS di Reggio Emilia - Presidio ospedaliero provinciale sede di Reggio Emilia, Reggio Emilia, Italy
- Netherlands (2):
  - Amphia Hospital, Breda
  - Reinier de Graaf Hospital, Delft
- United Kingdom (3):
  - Belfast Trust, City Hospital, Belfast
  - Guy's and St Thomas' Hospitals NHS Foundation Trust, London
  - King's College Hospital NHS Foundation, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Northouse LL, Mood DW, Schafenacker A, Kalemkerian G, Zalupski M, LoRusso P, Hayes DF, Hussain M, Ruckdeschel J, Fendrick AM, Trask PC, Ronis DL, Kershaw T. Randomized clinical trial of a brief and extensive dyadic intervention for advanced cancer patients and their family caregivers. Psychooncology. 2013 Mar;22(3):555-63. doi: 10.1002/pon.3036. Epub 2012 Jan 31. PMID 22290823
- [Background] Northouse L, Schafenacker A, Barr KL, Katapodi M, Yoon H, Brittain K, Song L, Ronis DL, An L. A tailored Web-based psychoeducational intervention for cancer patients and their family caregivers. Cancer Nurs. 2014 Sep-Oct;37(5):321-30. doi: 10.1097/NCC.0000000000000159. PMID 24945270
- [Background] Northouse L, Kershaw T, Mood D, Schafenacker A. Effects of a family intervention on the quality of life of women with recurrent breast cancer and their family caregivers. Psychooncology. 2005 Jun;14(6):478-91. doi: 10.1002/pon.871. PMID 15599947
- [Background] Larkin PJ, Dierckx de Casterle B, Schotsmans P. Multilingual translation issues in qualitative research: reflections on a metaphorical process. Qual Health Res. 2007 Apr;17(4):468-76. doi: 10.1177/1049732307299258. PMID 17416700
- [Derived] May P, Smith S, Jallow M, Kalinjuna T, De Vlemnick A, Matthys O, Van Goethem V, Groenvold M, Guerin S, Turola E, Bakker E, Brazil K, Harding R, Northouse L, Hudson P, Cohen J, Charles N; DIAdIC consortium. Assessing the cost-effectiveness of two psychoeducational interventions for people with cancer and their caregivers: An economic evaluation of the multi-country DIAdIC trial. Contemp Clin Trials. 2026 Jan 21:108240. doi: 10.1016/j.cct.2026.108240. Online ahead of print. PMID 41577124
- [Derived] De Vleminck A, Matthys O, Turola E, Dierickx S, Dombrecht L, Van Goethem V, Deliens L, Lapeire L, Hudson P, Eecloo K, Brazil K, Groenvold M, Di Leo S, van der Heide A, Normand C, Harding R, Pilch M, Northouse L; DIAdIC Team; Cohen J. Impact of a nurse-led and a web-based psychoeducational program for advanced cancer patients and their caregivers: Results of a three-arm randomized controlled trial. Int J Nurs Stud. 2025 Nov;171:105192. doi: 10.1016/j.ijnurstu.2025.105192. Epub 2025 Aug 19. PMID 40925214
- [Derived] Matthys O, De Vleminck A, Dierickx S, Deliens L, Van Goethem V, Lapeire L, Groenvold M, Lund L, Arnfeldt CM, Sengeloev L, Pappot H, Johnsen AT, Guerin S, Larkin PJ, Jordan C, Connolly M, D'Alton P, Costantini M, Di Leo S, Guberti M, Turola E, van der Heide A, Witkamp E, Rietjens J, van der Wel M, Brazil K, Prue G, Reid J, Scott D, Bristowe K, Harding R, Normand C, May P, Cronin C, Northouse L, Hudson P, Cohen J. Effectiveness of a nurse-delivered (FOCUS+) and a web-based (iFOCUS) psychoeducational intervention for people with advanced cancer and their family caregivers (DIAdIC): study protocol for an international randomized controlled trial. BMC Palliat Care. 2021 Dec 28;20(1):193. doi: 10.1186/s12904-021-00895-z. PMID 34963453